CLINICAL TRIAL: NCT01109056
Title: Safety and Efficacy of Cyclosporine Ophthalmic Emulsion in Patients With Primary Pterygium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192371-019
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-05

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cyclosporine ophthalmic emulsion 0.05% (Experimental): One drop in the study eye (or eyes) administered four times daily (QID)
  Interventions: Drug: cyclosporine ophthalmic emulsion 0.05%
- Vehicle (Placebo Comparator): One drop in the study eye (or eyes) administered four times daily (QID)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: cyclosporine ophthalmic emulsion 0.05% — One drop in the study eye (or eyes) administered four times daily (QID)
  Other Names: RESTASIS®
  Arms: cyclosporine ophthalmic emulsion 0.05%
Drug: Vehicle — One drop in the study eye (or eyes) administered four times daily (QID)
  Arms: Vehicle

SUMMARY:
This study will evaluate the safety and efficacy of Cyclosporine Ophthalmic Emulsion 0.05% (RESTASIS®) in patients with primary pterygium (abnormal growth on surface of eye).

ELIGIBILITY:
Inclusion Criteria:

* Have a pterygium in at least one eye that has not been previously removed with surgery

Exclusion Criteria:

* Uncontrolled systemic disease
* Active eye disease
* Current or anticipated use of topical eye medications other than artificial tears.
* Anticipated wearing of contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Glendale, California, United States
- Randwick, New South Wales, Australia
- Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclosporine Ophthalmic Emulsion 0.05% | Vehicle
Started | 57 | 58
Completed | 50 | 53
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine Ophthalmic Emulsion 0.05% | Vehicle | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Customized [Number; unit: Participants]
  <45 years | 13 | 15 | 28
  Between 45 and 65 years | 36 | 36 | 72
  >65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 41 | 35 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Pterygium Hyperemia Responders at Week 16
Description: Number of pterygium hyperemia responders at Week 16 as measured by the Pterygium Hyperemia Grading Scale. The Pterygium Hyperemia Grading Scale is a 6-point scale (0=absent, 1=trace, 2=mild, 3=moderate, 4=moderately severe, 5=severe). A responder is defined as a patient demonstrating at least a 2-grade decrease from baseline in pterygium hyperemia.
Time Frame: Week 16
Population: Modified Intent to Treat:
  All randomized patients who received study treatment and had a baseline and at least one post-baseline assessment of pterygium hyperemia
Measure: Number; unit: Participants
Arm/Group | Cyclosporine Ophthalmic Emulsion 0.05% | Vehicle
Number analyzed (Participants) | 56 | 57
Participants | 6 | 8

2. Primary Outcome: Change From Baseline in Severity Grade of Pterygium Hyperemia at Week 16
Description: Change from Baseline in Severity Grade of Pterygium Hyperemia at Week 16. The Pterygium Hyperemia Grading Scale is a 6-point scale (0=absent, 1=trace, 2=mild, 3=moderate, 4=moderately severe, 5=severe). A negative number change from baseline is an improvement and a positive number change from baseline is a worsening.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine Ophthalmic Emulsion 0.05% | Vehicle
Number analyzed (Participants) | 56 | 57
Scores on a Scale
  Baseline | 3.1 (0.35) | 3.2 (0.37)
  Change from Baseline at Week 16 | -0.7 (0.76) | -0.8 (0.75)

3. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index© (OSDI©) Questionnaire Score at Week 16
Description: Change from baseline in Ocular Surface Disease Index© (OSDI©) Questionnaire score at Week 16. The OSDI© is a 12-question survey for patients to document their dry eye disease symptoms. Each question is rated on a 5-point scale (0=none of the time and 4 = all of the time). The scores are totaled over the 12 questions and normalized/converted to a score of 0-100 (0=no disability and 100=complete disability). A negative number change from baseline represents an improvement.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cyclosporine Ophthalmic Emulsion 0.05% | Vehicle
Number analyzed (Participants) | 56 | 57
Scores on a Scale
  Baseline | 20.2 (16.97) | 29.3 (26.89)
  Change from Baseline at Week 16 | -3.1 (14.95) | -10.5 (16.02)

ADVERSE EVENTS:
Description: The Safety Population was used to calculate the number of participants at risk for SAEs and AEs, and is defined as all randomized and treated patients.
Arm/Group | Cyclosporine Ophthalmic Emulsion 0.05% | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/56 | 1/58
Other Adverse Events (participants affected / at risk) | 19/56 | 16/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cyclosporine Ophthalmic Emulsion 0.05% (N=56) | Vehicle (N=58)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/16 | 0/23
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cyclosporine Ophthalmic Emulsion 0.05% (N=56) | Vehicle (N=58)
Eye Irritation (Eye disorders) | 4 | 3
Conjunctival hyperaemia (Eye disorders) | 4 | 2
Eye Pain (Eye disorders) | 3 | 2
Instillation Site Pain (General disorders) | 3 | 2
Lacrimation Increased (Eye disorders) | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 7
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/16 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.